CLINICAL TRIAL: NCT05819736
Title: Pharmacokinetics Study Of Rivaroxaban and Apixaban in Cancer Patients
Acronym: EPRAPAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, Clinical Professor, Clinical Investigation Center Paris Est, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: 2022-10-15
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Anticoagulants and Thrombotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rivaroxaban: Cancer patients treated with rivaroxaban
  Interventions: Other: Monitoring
- Apixaban: Cancer patients treated with apixaban
  Interventions: Other: Monitoring

INTERVENTIONS:
Other: Monitoring — Monitoring

SUMMARY:
Direct oral anticoagulants (DOACs) are now recommended as a first-line option in cancer patients with venous thromboembolism or atrial fibrillation. However, current international clinical practice guidelines and product inserts suggest caution and/or avoidance in using DOACs in case of potential potential drug-drug interactions (DDI), including DDI with anticancer therapies. Indeed, potential important DDIs can affect the efficacy and safety of DOACs and/or anticancer therapies and/or other interfering medications in these patients. Data about the pharmacokinetics (PK) of DOACs in cancer patients are scarce. By using a PK approach, this study aims :

* to describe the PK profile of rivaroxaban and apixaban in adult cancer patients with venous thromboembolism or atrial fibrillation from a real-world setting
* to identify factors (age, weight, renal function, co-morbidities, etc) influencing the PK profile of rivaroxaban and apixaban in adult cancer with venous thromboembolism or atrial fibrillation from a real-world setting.

DETAILED DESCRIPTION:
Direct oral anticoagulants (DOACs) are now recommended as a first-line option in cancer patients with venous thromboembolism or atrial fibrillation. However, current international clinical practice guidelines and product inserts suggest caution and/or avoidance in using DOACs in case of potential potential drug-drug interactions (DDI), including DDI with anticancer therapies. Indeed, potential important DDIs can affect the efficacy and safety of DOACs and/or anticancer therapies and/or other interfering medications in these patients. Data about the pharmacokinetics (PK) of DOACs in cancer patients are scarce. By using a PK approach, this study aims :

* to describe the PK profile of rivaroxaban and apixaban in adult cancer patients with venous thromboembolism or atrial fibrillation from a real-world setting
* to identify factors (age, weight, renal function, co-morbidities, etc) influencing the PK profile of rivaroxaban and apixaban in adult cancer with venous thromboembolism or atrial fibrillation from a real-world setting

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with age ≥ 18 years
* Cancer (other than basal-cell or squamous-cell carcinoma of the skin), either active or diagnosed within 6 months prior to inclusion
* Confirmed symptomatic or venous thromboembolism or confirmed atrial fibrillation
* Patients affiliated with a health insurance system
* Able to provide written informed consent.

Exclusion Criteria:

* Age <18 years
* Pregnancy or breastfeeding
* Patients not affiliated with a health insurance system
* Patient subject to a measure of protection
* Legally protected adults
* Life expectancy < 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients with atrial fibrillation or venous thromboembolism receiving rivaroxaban or apixaban in a real-life clinical setting
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Population pharmacokinetic evaluation | 3 years
  Estimated area under the curve (AUC) of each of the 2 drugs studied

SECONDARY OUTCOMES:
Safety evaluation | 3 years
  Any thromboembolic event or major bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Blanchet, PharmD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Corinne Frere, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Centre d'Investigation Clinique Hôpital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided